CLINICAL TRIAL: NCT04583605
Title: Does PREVENA Vacuum-assisted Closure Reduce Lymphorrhoea Compared to Conventional Wound Closure After Axillary and Inguinal Lymph Node Dissection in the Management of Metastatic Cutaneous Skin Tumors ?
Brief Title: The Aim of This Study is to Demonstrat That Vacuum-assisted Closure Versus Conventional Wound Closure Enables to Diminish Local Complications After Lymph Node Dissection in Patients With Metastatic Skin Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: MR004
Record Dates: First submitted 2020-07-20; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-07

CONDITIONS: Melanoma; Skin Cancer; Epidermoid Carcinoma; Neuroendocrine Carcinoma; Lymph Node Metastases
Keywords: vacuum assisted closure; PRENEVA; lymph node dissection
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Neuroendocrine; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PREVENA: A vacuum wound closure therapy like PREVENA is applied after axillary or inguinal lymph node dissection in the management of metastatic skin tumors
  Interventions: Device: PREVENA
- NON PREVENA: A conventional wound closure is applied after axillary or inguinal lymph node dissection in the management of metastatic skin tumors

INTERVENTIONS:
Device: PREVENA — A negative pressure wound closure therapy is used after lymph node dissection
  Groups: PREVENA

SUMMARY:
In this study, we compared a negative pressure wound therapy, versus a conventional dressing in order to evaluate the most efficient wound therapy closure after axillary and inguinal lymph nodes dissections in the management of metastatic skin tumors. A vacuum assisted closure therapy should prevent these comorbidities.

DETAILED DESCRIPTION:
Lymphorrhoea, lymphedema and lymphocyte are significant and common complications after axillary and inguinal lymph nodes dissections. A vacuum assisted closure therapy should prevent these comorbidities. In this study, we compared PREVENA, a negative pressure wound therapy, versus conventional dressings. We evaluated the wound complications at the seventh day, the thirtieth day and at this end of the first year after surgery. It is a retrospective study of about ninety lymph nodes dissections among with there were seventy times the use of a negative pressure wound therapy, PREVENA.

ELIGIBILITY:
Inclusion Criteria:

* major patient affected by a metastatic skin tumors
* the primitive skin tumor is either a mélanoma, either squamous cell carcinoma , or a neuroendocrine tumor

Exclusion Criteria:

* lymph node dissection resumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major patient affected by a metastatic skin tumors
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Is there a visible scar disunion ? | between day 1 and day 7, between day 7 and day 30, between day 30 and first year end
  Yes if there is a scar opening, no if there isn't
Is there lymphorrhoea from the scar ? | between day 1 and day 7, between day 7 and day 30, between day 30 and first year end
  Yes if there is lymph coming from the the scar, no if there isn't.

SECONDARY OUTCOMES:
Are there lymphocele punctures ? | between day 1 and day 7, between day 7 and day 30, between day 30 and first year end
  Yes if there is any lymphocele puncture, no if there isn't
Is there any lymphoedema ? | between day 1 and day 7, between day 7 and day 30, between day 30 and first year end
  Yes if there is arm or leg lymphoedema, no if there isn't

CONTACTS AND LOCATIONS:
Overall Officials: Manuela PEREZ, Study Director — Visceral Surgery Department
Locations (1):
- CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Poirier A, Albuisson E, Bihain F, Granel-Brocard F, Perez M. Does Preventive Negative Pressure Wound Therapy (NPWT) reduce local complications following Lymph Node Dissection (LND) in the management of metastatic skin tumors? J Plast Reconstr Aesthet Surg. 2022 Dec;75(12):4403-4409. doi: 10.1016/j.bjps.2022.08.054. Epub 2022 Aug 24. PMID 36283927